CLINICAL TRIAL: NCT01323933
Title: A Phase 1, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AB0024 in Adult Patients With Advanced Solid Tumors
Brief Title: First-in-human Study of AB0024 to Evaluate Safety and Tolerability in Adults With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Zung Thai, MD/ Medical Monitor, Gilead Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB0024-101; NCT01158872 (obsolete NCT alias)
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Neoplasms
Keywords: Solid tumors; Oncology; Cancer
MeSH Terms: conditions — Neoplasms | interventions — simtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AB0024 (Experimental): The starting dose for Part A will be 1 mg/kg. Subsequent doses of 3, 10, and 20 mg/kg are planned. Three to 6 patients will be enrolled using a 3 + 3 design. Doses of AB0024 will be administered on Days 1, 15, 29, and 43 to characterize the safety, tolerability, and PK.
  The dose expansion phase of the study will begin upon completion of the dose escalation phase. Up to 20 patients will be enrolled into one or two cohorts of Part B. The first expansion cohort will be dosed up to the MTD defined as the highest dose level with an observed incidence of DLT in <33% of patients enrolled from Part A.
  Interventions: Drug: AB0024

INTERVENTIONS:
Drug: AB0024 — Comparison of different dosages of drug

SUMMARY:
Analysis of safety, tolerability, and PK data will provide information that will guide future development of AB0024.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, sequential dose escalation study to evaluate AB0024 in patients with advanced solid tumors. The study will consist of two parts: Part A will be a dose escalation, and Part B will be a dose expansion.The primary objective of this study is to characterize the safety, tolerability, and PK of AB0024 after multiple IV administrations in patients with advanced solid tumors. The secondary objectives are to measure the tumor response by modified RECIST and to evaluate the formation of anti-AB0024 antibodies.

Patients will receive infusions of AB0024 every two weeks. Patients will be seen weekly for safety assessments and collection of blood samples. Patients who do not show evidence of disease progression by clinical assessment or by CT or MRI may continue receiving AB0024 every 2 weeks until disease progression (clinical or radiographic), study drug intolerance, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced malignant solid tumor that is refractory to, intolerant of, or for which no standard of therapy is available
* Measurable or evaluable disease
* ECOG Performance Status of ≤2
* No known active central nervous system (CNS) tumors or CNS metastases
* Adequate organ function

Exclusion Criteria:

* Myocardial infarction within the last 6 months of study Day 1, symptomatic congestive heart failure (New York Heart Association Classification > Class II), unstable angina, or unstable cardiac arrhythmia requiring medication
* History of surgery within 28 days prior to enrollment or anticipated surgery during the study period
* Anti-tumor therapy (chemotherapy, antibody therapy, molecular targeted therapy, retinoid therapy, hormonal therapy) within 28 days of study Day 1 (six weeks for nitrosoureas, mitomycin C, antibodies, or molecular agents with t½ >10 days); (concurrent use of hormone therapy for breast or prostate cancer is permitted)
* Treatment with immune modulators including, but not limited to, cyclosporine and tacrolimus within two weeks prior to enrollment
* Concurrent or prior (within 30 days of study Day 1) anticoagulation therapy; (low-dose warfarin [<2 mg/day] for prophylaxis against central venous catheter thrombosis is allowed)
* Patient with tumor that is infiltrating or invading a major blood vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To characterize the safety, tolerability, and pharmacokinetics (PK) of AB0024 after multiple intravenous (IV) administrations in patients with advanced solid tumors. | Day 71

SECONDARY OUTCOMES:
To measure the tumor response by modified Response Evaluation Criteria in Solid Tumors (RECIST) and to evaluate the formation of anti-AB0024 antibodies. | Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Patricia LoRusso, DO, Principal Investigator — Barbara Ann Karmanos Cancer Institute; Anthony Tolcher, MD, Principal Investigator — South Texas Accelerated Research Therapeutics
Locations (2):
- United States (2):
  - Karmanos Cancer Institute, Detroit, Michigan
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

REFERENCES:
- [Derived] Barker HE, Cox TR, Erler JT. The rationale for targeting the LOX family in cancer. Nat Rev Cancer. 2012 Jul 19;12(8):540-52. doi: 10.1038/nrc3319. PMID 22810810